CLINICAL TRIAL: NCT00359866
Title: Pelvic IMRT With Tomotherapy: A Phase I Feasibility Study in Post-Hysterectomy Cervical Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 05-0977 / 201104019
Record Dates: First submitted 2006-08-02; First posted 2006-08-03 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Uterine Cervical Neoplasms
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pelvic IMRT with Tomotherapy (Experimental): Helical tomotherapy will be used to plan and deliver the radiation treatment.
  Treatment volume will include the upper third of the vagina and para-vaginal tissue and the common, external and internal iliac nodal regions.
  External beam radiation will be delivered in 160-180 cGy daily fractions to a total dose of 4500-5120 cGY.
  Receive treatment once a day for five days a week for approximately 6 weeks.
  Treating physician will make determination if patient is to receive intracavitary brachytherapy.
  Treating physician will make determination if patient is to receive chemotherapy (allowed but not mandated).
  Interventions: Radiation: IMRT with tomotherapy

INTERVENTIONS:
Radiation: IMRT with tomotherapy

SUMMARY:
Indications for post-hysterectomy radiation therapy (RT) have been well established by clinical data. Adjuvant RT has demonstrated local control and survival benefit. In patients with nodal disease, adjuvant chemotherapy concurrent with radiation has further improved the clinical outcome. The acute hematological and gastrointestinal toxicity of concurrent chemo-radiotherapy can be quite high, sometimes preventing patients from completed their full treatment course, potentially compromising the therapeutic benefit of treatment. Intensity modulated radiation therapy (IMRT) is an advanced method of delivering external beam radiation that may minimize the volume of normal tissue irradiated to high dose and thus decrease the risk of normal tissue toxicity. Helical tomotherapy is a novel treatment device with sophisticated imaging and treatment delivery features that are optimally suited for IMRT. There are retrospective clinical data supporting the use of non-tomotherapy delivered IMRT to treat patients with gynecologic cancers. The proposed study will prospectively test whether helical tomotherapy is a feasible method for delivering IMRT in post-hysterectomy cervical cancer patients receiving adjuvant RT. Here, the question of feasibility is simply one of verifying that target volumes are reliably covered by 'sculpted' IMRT high-dose regions. Although this is not a treatment effectiveness study, we will also follow the clinical outcome of these patients, including toxicity, local control and survival, in anticipation that this information will be valuable if the treatment modality is judged feasible and will be used for further treatments of this patient population.

DETAILED DESCRIPTION:
Patients with cervical cancer receiving post-operative radiotherapy (RT) for high risk features found on pathologic review will be treated with pelvic intensity modulated radiation therapy (IMRT). Helical tomotherapy will be used to plan and deliver the radiation treatment. Treatment volume will include the upper third of the vagina and para-vaginal tissue and the common, external and internal iliac nodal regions. External beam radiation will be delivered in 180 cGy daily fractions to a total dose of 5040 cGy. Patients will receive once a day treatment five days a week, for approximately 6 weeks. Concurrent chemotherapy and/or intracavitary brachytherapy may be included in the treatment plan at the discretion of the treating physician, consistent with routine clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18
* Karnofsky Performance Status of >= 60
* FIGO Stage I -IIB
* Pathologic confirmation of cervical cancer
* Status post hysterectomy
* Patients with local or regional metastases are eligible for this protocol, but not those with distant metastases

Exclusion Criteria:

* Age < 18
* Karnofsky Performance Status < 60
* Radiographic or pathologic evidence of distant metastatic disease
* Prior pelvic radiation therapy, other than trans-vaginal ring brachytherapy irradiation for acute hemostasis

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2006-02; Primary Completion 2010-07 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Determine the feasibility of using helical tomotherapy to deliver IMRT | After all patients are enrolled and complete treatment
  Feasibility is defined as the ability to deliver 95% of the prescription dose to 90% of the original planning target volume in at least 90% of the patients, as verified by actual dose delivered calculations using on board CT scan.

SECONDARY OUTCOMES:
Measure the acute toxicity | Up through 30 days after completion of treatment
Measure the late toxicity | Starting 30 days from completion of treatment through 1 year post start of treatment
Measure the local, regional, and distant recurrence rates | 5 years after completion of treatment
Measure the 5-year disease free and 5-year overall survival rates | 5 years after completion of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Perry W Grigsby, M.D., Principal Investigator — Washington University Medical School
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu